CLINICAL TRIAL: NCT06547918
Title: Safety and Effectiveness of the Omnipod® 5 SmartAdjust 2.0 System in Individuals With Type 1 and Type 2 Diabetes
Brief Title: SmartAdjust 2.0 System With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA2.0 Feasibility (NZ)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus
Keywords: Type 1 Diabetes T1D; Type 2 Diabetes T2D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Participants with Type 1 and Type 2 diabetes (Experimental)
  Interventions: Device: Omnipod 5 SA2.0 System

INTERVENTIONS:
Device: Omnipod 5 SA2.0 System — The Omnipod 5 SA2.0 System provides automated insulin delivery based on Continuous Glucose Monitoring (CGM) values.

SUMMARY:
This study will evaluate the safety and effectiveness of the Omnipod 5 SmartAdjust 2.0 System in individuals aged 2-70 years with type 1 or type 2 diabetes.

DETAILED DESCRIPTION:
This is a single-arm study that will enroll up to 75 participants aged 2-70 years with Type 1 diabetes and aged 16-70 years with Type 2 diabetes in order to have a minimum of 48 participants (24 with Type 1 Diabetes and 24 with Type 2 Diabetes) initiate the use of the Omnipod 5 SA2.0 System.

The Study will take part in two periods. Participants who do not have the minimum requirement of CGM data will undergo 2 weeks of Standard Therapy while using a Dexcom G6 in an outpatient setting before proceeding to Period 1.

During period 1, all participants will use the Omnipod SmartAdjust 2.0 System in an outpatient setting for up to six weeks. Period 2 is an optional extension of time that allows participants to continue using the Omnipod 2.0 SmartAdjust System for an additional six months.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all the following criteria at screening to be included in the study:

1. Age at time of consent 2-70 years (inclusive)
2. Diabetes diagnosis, based on Investigator's clinical judgement, and meets the following:

   * Type 1 Diabetes: 2-70 years old with A1c <11%. Diagnosed for at least 6 months for participants aged 2- <7 years or at least 1 year for participants aged 7-70 years. OR
   * Type 2 Diabetes: 16-70 years old, diagnosed with T2D and on current insulin regimen for at least 3 months. Includes basal-bolus, pre-mix, or basal only users. For basal-bolus and premix users, must have A1c < 12.0%. For basal only users must have A1c > 7.0% and < 12.0%.
3. Living with a parent or guardian if < 16 years old
4. Currently using U-100 rapid-acting insulin analogs with insulin pump or basal-bolus, pre-mix, or basal only users suitable for conversion to pump therapy for at least 3 months prior to study start
5. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novorapid, or their generic equivalents
6. Deemed appropriate for pump therapy per Investigator's assessment considering previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
7. Stable doses over the preceding 4 weeks of other glucose-lowering medications, as determined by Investigator, including within class dose equivalent medication
8. Stable doses over the preceding 4 weeks of weight loss medications that may affect glycemic control directly and/or indirectly, as determined by Investigator
9. Investigator has confidence that the participant and/or caregiver can safely operate all study devices and can adhere to the protocol
10. Willing to wear the system, including Pods, continuously throughout the study
11. If female of childbearing potential, willing and able to have pregnancy testing

Exclusion Criteria:

Individuals who meet any of the following criteria at screening will be excluded from study participation:

1. Any medical condition, which in the opinion of the Investigator, would put the participant at an unacceptable safety risk
2. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the 12 months prior to screening
3. Any planned surgery during the study which could be considered major in the opinion of the Investigator
4. Severe retinopathy based on retinal screening performed within the last 24 months
5. History of severe hypoglycemia in the past 6 months. Severe hypoglycemia is defined as an event that requires the assistance of another person due to altered consciousness, and requires another person to actively administer carbohydrate, glucagon, or other resuscitative actions
6. History of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS) in the past 6 months, unrelated to an intercurrent illness or infusion failure
7. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
8. Blood disorder or dyscrasia within 3 months prior to screening, including use of hydroxyurea, which in the Investigator's opinion could interfere with determination of HbA1c
9. Plans to receive blood transfusion over the course of the study
10. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilization such as tubal ligation or hysterectomy, or vasectomized partner)
11. Participation in another clinical study using an investigational drug or device within 30-days or intends to participate in any other study during this study period
12. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the Investigator's clinical judgment
13. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member of any of the aforementioned

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range <3.9 mmol/L (<70 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 and Period 2 (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time in hyperglycemic range >13.9 mmol/L (>250 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)

SECONDARY OUTCOMES:
Mean glucose (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time < 3.0 mmol/L (<54 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time > 10.0 mmol/L (>180 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time > 16.7 mmol/L (>300 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time between 3.9-10.0 mmol/L (70-180 mg/dL) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from study provided continuous glucose monitor (CGM)
Standard deviation (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from the continuous glucose monitor (CGM)-measured glucose variability with the standard deviation (SD)
Coefficient of variation (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Glucose metric from the continuous glucose monitor (CGM)-measured glucose variability with the coefficient of variation (CV)
Average total daily insulin (TDI) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Measure of insulin requirements
Average TDI/kg (assessed by diabetes type (type 1 and type 2)) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to Standard Therapy
  Measure of insulin requirements
Incidence rate of severe hypoglycemia (events per person months) (assessed by diabetes type (type 1 and type 2)) | End of Period 1 upto 6 weeks and Period 2 upto 6 months (optional) compared to participant reported events over the preceding year prior to Visit 4
  Measure of insulin requirements
Incidence rate of diabetic ketoacidosis (DKA) and/or hyperosmolar (assessed by diabetes type (type 1 and type 2)) hyperglycemic state (HHS) (events per person months) | End of Period 1 which is upto 6 weeks and Period 2 which is upto 6 months (optional) compared to participant reported events over the preceding year prior to Visit 4
  Measure of insulin requirements

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - University of Otago, Christchurch, Christchurch
  - Wellington Regional Hospital, Wellington